CLINICAL TRIAL: NCT03647475
Title: Onyx ONE Clear: A Single Arm Trial With Resolute Onyx in ONE-Month DAPT for High-Bleeding Risk Patients Who Are Considered One-Month Clear (Onyx ONE Clear)
Brief Title: A Single Arm Trial With Resolute Onyx in ONE-Month DAPT for High-Bleeding Risk Patients Who Are Considered One-Month Clear (Onyx ONE Clear)
Acronym: Onyx ONE Clear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT18015RES008
Record Dates: First submitted 2018-08-17; First posted 2018-08-27 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, single arm trial enrolling eligible subjects in the United States and Japan. Subjects will remain in the study with follow-up clinical assessments through 2 years, study exit, or death, whichever comes first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent (Experimental): Subjects who fulfilled the inclusion criteria and none of the exclusion criteria were treated with a Resolute Onyx stent followed by one-month DAPT. The clinical safety of the Resolute Onyx stent as compared to a performance goal was evaluated using a composite safety endpoint of cardiac death and myocardial infarction at 1 year for a one-month clear population.
  Interventions: Combination Product: Device: Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System Treatment Followed by one-month DAPT

INTERVENTIONS:
Combination Product: Device: Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System Treatment Followed by one-month DAPT — To evaluate the clinical safety of the Resolute Onyx stent with use of one-month DAPT in subjects deemed at high risk for bleeding and/or medically unsuitable for more than one-month DAPT treatment.

SUMMARY:
The purpose of this trial is to evaluate the clinical safety and effectiveness of the Resolute Onyx stent in subjects deemed at high risk for bleeding and/or medically unsuitable for more than 1 month DAPT treatment receiving reduced duration (1 month) of DAPT following stent implantation.

ELIGIBILITY:
Inclusion Criteria:

To qualify as high-bleeding risk and/or a candidate for 1-month DAPT, subject had to meet at least one of the criteria detailed below:

* Adjunctive chronic oral anticoagulation treatment planned to continue after PCI
* Age ≥ 75 years old
* Baseline Hgb <11 g/dl (or anemia requiring transfusion during the 4 weeks prior to procedure)
* Any prior documented intracerebral bleed
* Any documented stroke in the last 12 months
* Hospital admission for bleeding during the prior 12 months
* Active non-skin cancer currently undergoing treatment or surveillance (in lieu of treatment)
* Planned daily NSAID (other than aspirin) or steroids for ≥30 days after PCI
* Planned surgery that would require interruption of DAPT (within the next 12 months)
* Renal failure defined as: Creatinine clearance <40 ml/min
* Thrombocytopenia (PLT <100,000/mm3)
* Severe chronic liver disease defined as: subjects who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice
* Expected non-compliance for at least 6 months DAPT for other medical reasons

Exclusion Criteria:

* Pregnant and breastfeeding women
* Subjects requiring a planned PCI procedure after 1 month of index procedure
* Procedure planned to require non-trial stents, stand-alone POBA, or stand-alone atherectomy
* Active bleeding at the time of inclusion
* Cardiogenic shock
* Subject with planned surgery or procedure necessitating discontinuation of DAPT within one month following index procedure
* Subject not expected to comply with long-term single antiplatelet therapy
* A known hypersensitivity or contraindication to aspirin, heparin and bivalirudin, P2Y12 inhibitors, mTOR inhibiting drugs such as zotarolimus, Biolimus A9 (or its derivatives), cobalt, nickel, platinum, iridium, chromium, molybdenum, polymer coatings (eg, BioLinx™), stainless steel (or other metal ions found in 316L stainless steel), zinc, or a sensitivity to contrast media, which cannot be adequately pre-medicated.
* PCI during the previous 6 months for a lesion other than the target lesion of the index procedure
* Participation in another clinical study within 12 months after index procedure
* Subjects with life expectancy of less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Atlanta Hospital, Atlanta, GA; Ajay Kirtane, MD, Principal Investigator — New York-Presbyterian Hospital/Columbia University Medical Center, New York, NY
Locations (4):
- United States (4):
  - Saint Joseph's Hospital Health Center, East Syracuse, New York
  - New York- Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - AnMed Health Medical Center, Anderson, South Carolina
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kandzari DE, Kirtane AJ, Windecker S, Latib A, Kedhi E, Mehran R, Price MJ, Abizaid A, Simon DI, Worthley SG, Zaman A, Choi JW, Caputo R, Kanitkar M, McLaurin B, Potluri S, Smith T, Spriggs D, Tolleson T, Nazif T, Parke M, Lee LC, Lung TH, Stone GW; Onyx ONE US/Japan Investigators. One-Month Dual Antiplatelet Therapy Following Percutaneous Coronary Intervention With Zotarolimus-Eluting Stents in High-Bleeding-Risk Patients. Circ Cardiovasc Interv. 2020 Nov;13(11):e009565. doi: 10.1161/CIRCINTERVENTIONS.120.009565. Epub 2020 Nov 10. PMID 33167705
- [Derived] Kang J, Abdul Ghapar AK, Selvaraj K, Hur SH, Tam CC, Jang Y, Chae IH, Kandzari DE, Kirtane AJ, Latib A, Kedhi E, Lung TH, You SJ, Windecker S, Stone GW, Kim HS. One-Month Dual Antiplatelet Therapy in High Bleeding Risk Asian Patients Undergoing Percutaneous Coronary Intervention - Onyx ONE Clear 2-Year Results. Circ Rep. 2024 Jul 6;6(8):333-340. doi: 10.1253/circrep.CR-24-0037. eCollection 2024 Aug 9. PMID 39132335
- [Derived] Toth GG, Kandzari DE, Kirtane AJ, Windecker S, Latib A, Kedhi E, Mehran R, Price MJ, Choi JW, Caputo R, Troquay R, Diderholm E, Singh S, Brar SS, Loussararian A, Chetcuti S, Tulli M, Stone GW, Lung TH, Mylotte D. Two-year results from Onyx ONE clear in patients with high bleeding risk on one-month DAPT with and without intracoronary imaging. Cardiovasc Revasc Med. 2024 Jan;58:60-67. doi: 10.1016/j.carrev.2023.07.016. Epub 2023 Jul 24. PMID 37550123

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, the 752 subjects enrolled in the US & Japan were pooled with A Randomized Controlled Trial With Resolute Onyx in One Month Dual Antiplatelet Therapy (DAPT) for High-Bleeding Risk Patients" (NCT03344653). Subjects enrolled under NCT03344653 were in regions outside of the US and Japan.
Period: Overall Study
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Started | 752
NCT03647475 - Included in One Month Clear Analysis Population | 601
NCT03344653- Included in One Month Clear Analysis Population | 905
Completed | 75
Not Completed | 677

BASELINE CHARACTERISTICS:
Population: The analysis population combines eligible subjects enrolled in the Onyx ONE US & Japan Trial (NCT03647475) and Onyx ONE Global RCT (NCT03344653) who received the Resolute Onyx stent only, were adherent to DAPT for the one-month period, were event-free on or prior to the DAPT stop date, and transitioned from DAPT to SAPT one month after procedure.
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 241
  >=65 years | 1265
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 487
  Male | 1019
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 564
  Japan | 37
  Australia | 85
  Austria | 11
  Belgium | 27
  Bulgaria | 52
  France | 12
  Hong Kong | 20
  Ireland | 27
  Italy | 61
  Latvia | 11
  Lithuania | 6
  Malaysia | 100
  Netherlands | 50
  New Zealand | 33
  Norway | 2
  Poland | 23
  Singapore | 8
  Slovakia | 92
  Spain | 98
  Sweden | 25
  Switzerland | 12
  Thailand | 1
  United Kingdom | 43
  South Korea | 106

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint: Number of Participants With Cardiac Death and Myocardial Infarction
Description: Composite of cardiac death and myocardial infarction at one year for a one-month clear population [Time Frame: One month to one year]
Time Frame: One Month to one year
Population: The analysis population combines eligible subjects enrolled in the Onyx ONE US & Japan Trial (NCT03647475) and Onyx ONE Global RCT (NCT03344653) who received the Resolute Onyx stent only, and met the trial definition for one- month clear.
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 104

2. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: Defined as cardiac death, target vessel myocardial infarction (Q wave and non Q wave), or clinically driven target lesion revascularization(TLR) by percutaneous or surgical method
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 121

3. Secondary Outcome: Number of Participants With Procedure Success
Description: Attainment of <30% residual stenosis by QCA (or <20% by visual assessment) AND TIMI flow 3 after the procedure, using any percutaneous method without the occurrence of MACE during the hospital stay.
Time Frame: Procedure to hospital discharge, an average of 1.3 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 1295

4. Secondary Outcome: All Participants Deaths Including Cardiac Death
Description: All participants deaths including cardiac death
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 89

5. Secondary Outcome: Number of Patients With Major Cardiac Event
Description: Major adverse cardiac event (MACE) defined as composite of death, myocardial infarction, or repeat target lesion revascularization (clinically driven) by percutaneous or surgical methods
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 174

6. Secondary Outcome: Number of Patients With Myocardial Infarction
Description: All myocardial infarction including Target Vessel Myocardial Infarction (TVMI)
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 72

7. Secondary Outcome: Number of Patients With Target Vessel Failure
Description: Target vessel failure (TVF) defined as composite of cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization (TVR) by percutaneous or surgical methods.
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 131

8. Secondary Outcome: Number of Patients With Revascularization
Description: All revascularizations (TLR, TVR and non-TVR)
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 84

9. Secondary Outcome: Number of Patients With Stent Thrombosis
Description: Stent thrombosis (per Academic Research Consortium (ARC) definition)
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 10

10. Secondary Outcome: Number of Patients With Bleeding
Description: Bleeding per BARC (Bleeding Academic Research Consortium) criteria. This criteria classifies bleeding events with BARC 1 being the least severe and type 5 being the most severe.
  Grouping of BARC categories:
  * BARC 3 to 5 - This included all bleeding events in BARC 3 to BARC 5 categories
  * BARC 2 to 5- This included all bleeding events in BARC 2 to BARC 5 categories
  * All BARC- This included all bleeding events BARC 1 through BARC 5
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants
  All BARC | 195
  BARC 3 to 5 | 60
  BARC 2 to 5 | 175

11. Secondary Outcome: Number of Patients With Stroke
Description: Stroke
Time Frame: One Month to One Year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Participants | 22

12. Secondary Outcome: Lesion Success
Description: The attainment of <30% residual stenosis by QCA (or < 20% by visual assessment) AND TIMI flow 3 after the procedure, using any percutaneous method
Time Frame: End of Procedure, an average of 42 minutes
Population: as for outcome 1
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Number analyzed (Lesions) | 1960
Lesions | 1817

13. Secondary Outcome: Device Success
Description: Attainment of <30% residual stenosis by QCA (or <20% by visual assessment) AND TIMI flow 3 after the procedure, using the assigned device only.
Time Frame: End of Procedure an average of 42 minutes
Population: as for outcome 1
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 1506
Number analyzed (Lesions) | 1960
Lesions | 1790

ADVERSE EVENTS:
Time Frame: From One Month to 365 Days
Description: For the purpose of this clinical investigation, reportable events ( Subjects enrolled in NCT03344653 and those enrolling in Japan were required to report all AEs per local regulations) in the subject population being evaluated were those that met the criteria for a Serious Adverse Event (SAE) and any AE related to the trial end points, including all bleeding events. For the purposes of the primary endpoint evaluation, events assessed from one month to 365 days were included in the analysis.
Arm/Group | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent
All-Cause Mortality (participants affected / at risk) | 89/1506
Serious Adverse Events (participants affected / at risk) | 591/1506
Other Adverse Events (participants affected / at risk) | 755/1506
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent (N=1506)
Anaemia (Blood and lymphatic system disorders) | 34 (38)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 7 (7)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 2 (2)
Normocytic Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Acute Coronary Syndrome (Cardiac disorders) | 8 (9)
Acute Left Ventricular Failure (Cardiac disorders) | 5 (5)
Acute Myocardial Infarction (Cardiac disorders) | 38 (40)
Angina Pectoris (Cardiac disorders) | 26 (26)
Angina Unstable (Cardiac disorders) | 16 (16)
Anginal Equivalent (Cardiac disorders) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 48 (59)
Atrial Flutter (Cardiac disorders) | 8 (8)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 2 (2)
Atrioventricular Block Complete (Cardiac disorders) | 5 (5)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1)
Atrioventricular Block Second Degree (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 8 (8)
Bundle Branch Block Left (Cardiac disorders) | 1 (1)
Bundle Branch Block Right (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 6 (6)
Cardiac Asthma (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 21 (22)
Cardiac Failure Acute (Cardiac disorders) | 8 (9)
Cardiac Failure Chronic (Cardiac disorders) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 40 (52)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2)
Chronic Left Ventricular Failure (Cardiac disorders) | 1 (1)
Conduction Disorder (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 14 (15)
Coronary Artery Dissection (Cardiac disorders) | 3 (3)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 7 (7)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1)
Coronary Ostial Stenosis (Cardiac disorders) | 2 (2)
Dressler's Syndrome (Cardiac disorders) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 4 (4)
Microvascular Coronary Artery Disease (Cardiac disorders) | 1 (1)
Mitral Valve Disease (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 2 (2)
Myocardial Haemorrhage (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 12 (12)
Myocardial Ischaemia (Cardiac disorders) | 7 (7)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Prosthetic Cardiac Valve Thrombosis (Cardiac disorders) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 7 (7)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 5 (5)
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 2 (2)
Haemorrhagic Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1)
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Vestibular Disorder (Ear and labyrinth disorders) | 1 (1)
Blindness Unilateral (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 5 (6)
Diabetic Retinopathy (Eye disorders) | 1 (1)
Eye Ulcer (Eye disorders) | 1 (1)
Macular Degeneration (Eye disorders) | 1 (1)
Retinal Artery Occlusion (Eye disorders) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Chronic Gastritis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Crohn's Disease (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Diverticulum (Gastrointestinal disorders) | 3 (3)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (3)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Erosive Duodenitis (Gastrointestinal disorders) | 1 (1)
Femoral Hernia (Gastrointestinal disorders) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1)
Gastric Perforation (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Erosion (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 12 (12)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhagic Ascites (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1)
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 4 (4)
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 2 (2)
Large Intestine Polyp (Gastrointestinal disorders) | 3 (3)
Levator Syndrome (Gastrointestinal disorders) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 (9)
Melaena (Gastrointestinal disorders) | 1 (1)
Mesenteric Artery Stenosis (Gastrointestinal disorders) | 1 (1)
Mouth Haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1)
Pharyngo-Oesophageal Diverticulum (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Tooth Impacted (Gastrointestinal disorders) | 1 (2)
Umbilical Hernia (Gastrointestinal disorders) | 4 (4)
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Varices Oesophageal (Gastrointestinal disorders) | 1 (1)
Adverse Drug Reaction (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (2)
Catheter Site Haemorrhage (General disorders) | 2 (2)
Chest Pain (General disorders) | 17 (18)
Death (General disorders) | 15 (15)
Fatigue (General disorders) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1)
Generalised Oedema (General disorders) | 1 (1)
Impaired Healing (General disorders) | 3 (3)
Implant Site Haemorrhage (General disorders) | 1 (1)
Incarcerated Hernia (General disorders) | 1 (1)
Infusion Site Extravasation (General disorders) | 1 (1)
Injection Site Extravasation (General disorders) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 18 (19)
Oedema Peripheral (General disorders) | 1 (1)
Peripheral Swelling (General disorders) | 1 (1)
Physical Deconditioning (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Sudden Cardiac Death (General disorders) | 4 (4)
Sudden Death (General disorders) | 2 (2)
Vascular Stent Stenosis (General disorders) | 22 (22)
Vascular Stent Thrombosis (General disorders) | 5 (5)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1)
Biliary Colic (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 2 (2)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 2 (2)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic Mass (Hepatobiliary disorders) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 1 (1)
Non-Alcoholic Steatohepatitis (Hepatobiliary disorders) | 1 (1)
Food Allergy (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Primary Amyloidosis (Immune system disorders) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 1 (1)
Abscess Jaw (Infections and infestations) | 1 (1)
Abscess Limb (Infections and infestations) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial Parotitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Bronchitis Viral (Infections and infestations) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 8 (9)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1)
Clostridium Difficile Infection (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Cytomegalovirus Oesophagitis (Infections and infestations) | 1 (1)
Dengue Fever (Infections and infestations) | 1 (1)
Device Related Infection (Infections and infestations) | 2 (2)
Device Related Sepsis (Infections and infestations) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 1 (1)
Diarrhoea Infectious (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Diverticulitis Intestinal Haemorrhagic (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Endocarditis Bacterial (Infections and infestations) | 1 (1)
Endocarditis Enterococcal (Infections and infestations) | 1 (1)
Enterococcal Bacteraemia (Infections and infestations) | 1 (1)
Enterocolitis Fungal (Infections and infestations) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 2 (3)
Gastroenteritis (Infections and infestations) | 6 (6)
Gastrointestinal Infection (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Infected Seroma (Infections and infestations) | 1 (1)
Infected Skin Ulcer (Infections and infestations) | 2 (2)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 3 (3)
Nosocomial Infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 43 (48)
Pneumonia Bacterial (Infections and infestations) | 4 (4)
Pneumonia Klebsiella (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 3 (3)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Renal Cyst Infection (Infections and infestations) | 1 (2)
Respiratory Tract Infection (Infections and infestations) | 5 (6)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 15 (16)
Septic Shock (Infections and infestations) | 2 (2)
Staphylococcal Bacteraemia (Infections and infestations) | 2 (2)
Streptococcal Bacteraemia (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 20 (23)
Urinary Tract Infection Bacterial (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 4 (4)
Wound Infection (Infections and infestations) | 1 (1)
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 3 (3)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Valve Replacement Complication (Injury, poisoning and procedural complications) | 1 (1)
Chemical Peritonitis (Injury, poisoning and procedural complications) | 1 (1)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 2 (2)
Costal Cartilage Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 4 (4)
Flail Chest (Injury, poisoning and procedural complications) | 1 (1)
Haemodialysis Complication (Injury, poisoning and procedural complications) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 3 (3)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Postoperative Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural Dizziness (Injury, poisoning and procedural complications) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Pulmonary Contusion (Injury, poisoning and procedural complications) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 2 (2)
Rib Fracture (Injury, poisoning and procedural complications) | 3 (3)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 4 (4)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 2 (2)
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Urinary Tract Stoma Complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood Glucose Fluctuation (Investigations) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1)
Cardiac Output Decreased (Investigations) | 1 (1)
Ejection Fraction Decreased (Investigations) | 3 (3)
Haemoglobin Decreased (Investigations) | 3 (3)
Heparin-Induced Thrombocytopenia Test Positive (Investigations) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1)
Pulmonary Function Test Decreased (Investigations) | 1 (1)
Stress Echocardiogram Abnormal (Investigations) | 1 (1)
Alcoholic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 (2)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Mineral Deficiency (Metabolism and nutrition disorders) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Wall Haematoma (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Haematoma Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 2 (2)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Atypical Fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Bone Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hypopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's Lymphoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered State Of Consciousness (Nervous system disorders) | 1 (1)
Amputation Stump Pain (Nervous system disorders) | 1 (1)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 3 (3)
Cerebral Infarction (Nervous system disorders) | 3 (3)
Cerebrovascular Accident (Nervous system disorders) | 10 (11)
Cerebrovascular Insufficiency (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Embolic Stroke (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Frontotemporal Dementia (Nervous system disorders) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 2 (2)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 3 (9)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 4 (4)
Lethargy (Nervous system disorders) | 2 (2)
Loss Of Consciousness (Nervous system disorders) | 2 (2)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 2 (2)
Myelopathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3)
Sciatica (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 3 (3)
Stupor (Nervous system disorders) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 11 (12)
Transient Global Amnesia (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 7 (7)
Vertebrobasilar Stroke (Nervous system disorders) | 1 (1)
Device Capturing Issue (Product Issues) | 1 (1)
Device Deposit Issue (Product Issues) | 1 (1)
Device Inappropriate Shock Delivery (Product Issues) | 1 (1)
Device Loosening (Product Issues) | 1 (1)
Device Malfunction (Product Issues) | 1 (1)
Lead Dislodgement (Product Issues) | 2 (2)
Stent Malfunction (Product Issues) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 (3)
Delirium (Psychiatric disorders) | 2 (2)
Dissociative Amnesia (Psychiatric disorders) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 30 (34)
Azotaemia (Renal and urinary disorders) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 2 (2)
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
End Stage Renal Disease (Renal and urinary disorders) | 6 (8)
Haematuria (Renal and urinary disorders) | 11 (11)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Nephropathy Toxic (Renal and urinary disorders) | 1 (1)
Renal Cyst Haemorrhage (Renal and urinary disorders) | 1 (2)
Renal Failure (Renal and urinary disorders) | 4 (4)
Renal Haematoma (Renal and urinary disorders) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 4 (4)
Ureterolithiasis (Renal and urinary disorders) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 9 (11)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 3 (3)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mediastinal Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Colostomy (Surgical and medical procedures) | 1 (1)
Hernia Repair (Surgical and medical procedures) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 1 (1)
Toe Operation (Surgical and medical procedures) | 1 (2)
Aortic Aneurysm (Vascular disorders) | 4 (4)
Aortic Dissection (Vascular disorders) | 1 (1)
Aortic Stenosis (Vascular disorders) | 12 (12)
Arteriosclerosis (Vascular disorders) | 1 (1)
Bleeding Varicose Vein (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 5 (5)
Dry Gangrene (Vascular disorders) | 2 (3)
Embolism Venous (Vascular disorders) | 1 (1)
Extremity Necrosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 3 (3)
Haemodynamic Instability (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 9 (10)
Hypertensive Crisis (Vascular disorders) | 4 (4)
Hypertensive Emergency (Vascular disorders) | 3 (3)
Hypertensive Urgency (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 7 (8)
Hypovolaemic Shock (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 3 (3)
Orthostatic Hypotension (Vascular disorders) | 2 (2)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 6 (6)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1)
Peripheral Artery Occlusion (Vascular disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 6 (7)
Peripheral Vascular Disorder (Vascular disorders) | 7 (7)
Steal Syndrome (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Vena Cava Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent (N=1506)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Anaemia Folate Deficiency (Blood and lymphatic system disorders) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic Disorder (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Schistocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3)
Angina Pectoris (Cardiac disorders) | 29 (32)
Angina Unstable (Cardiac disorders) | 2 (2)
Anginal Equivalent (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 14 (14)
Atrial Flutter (Cardiac disorders) | 2 (2)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Atrioventricular Block First Degree (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 3 (3)
Bundle Branch Block Left (Cardiac disorders) | 1 (1)
Bundle Branch Block Right (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 9 (9)
Cardiac Failure Chronic (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardiac Valve Disease (Cardiac disorders) | 1 (1)
Defect Conduction Intraventricular (Cardiac disorders) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vertigo Positional (Ear and labyrinth disorders) | 2 (2)
Cataract (Eye disorders) | 2 (2)
Conjunctival Haemorrhage (Eye disorders) | 4 (5)
Diplopia (Eye disorders) | 1 (1)
Eye Haemorrhage (Eye disorders) | 1 (1)
Eye Pain (Eye disorders) | 1 (1)
Lacrimation Increased (Eye disorders) | 1 (1)
Vitreous Haemorrhage (Eye disorders) | 1 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 6 (6)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3)
Anal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Anal Stenosis (Gastrointestinal disorders) | 1 (1)
Appendicolith (Gastrointestinal disorders) | 1 (1)
Atrophic Glossitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (4)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Gingival Hypertrophy (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6)
Rectal Haemorrhage (Gastrointestinal disorders) | 5 (5)
Tongue Disorder (Gastrointestinal disorders) | 1 (1)
Tongue Haemorrhage (Gastrointestinal disorders) | 3 (4)
Toothache (Gastrointestinal disorders) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Adverse Drug Reaction (General disorders) | 2 (2)
Asthenia (General disorders) | 2 (2)
Catheter Site Haematoma (General disorders) | 1 (1)
Catheter Site Haemorrhage (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 9 (9)
Chest Pain (General disorders) | 28 (28)
Drug Intolerance (General disorders) | 1 (1)
Exercise Tolerance Decreased (General disorders) | 1 (1)
Fatigue (General disorders) | 8 (8)
Hangover (General disorders) | 1 (1)
Malaise (General disorders) | 2 (3)
Non-Cardiac Chest Pain (General disorders) | 21 (22)
Oedema Peripheral (General disorders) | 7 (7)
Pain (General disorders) | 1 (1)
Peripheral Swelling (General disorders) | 2 (2)
Puncture Site Haematoma (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Biliary Colic (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic Lesion (Hepatobiliary disorders) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 1 (1)
Nonalcoholic Fatty Liver Disease (Hepatobiliary disorders) | 1 (1)
Contrast Media Allergy (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Cellulitis (Infections and infestations) | 5 (6)
Chronic Hepatitis C (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1)
Fungal Skin Infection (Infections and infestations) | 1 (2)
Furuncle (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 1 (1)
Helicobacter Infection (Infections and infestations) | 1 (1)
Infected Skin Ulcer (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Necrotising Soft Tissue Infection (Infections and infestations) | 1 (1)
Oral Candidiasis (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 5 (5)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 10 (10)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1)
Wound Sepsis (Infections and infestations) | 1 (1)
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous Graft Site Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 16 (19)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 2 (2)
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 3 (3)
Muscle Injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 2 (2)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1)
Periorbital Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Plaque Shift (Injury, poisoning and procedural complications) | 1 (2)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Hypertension (Injury, poisoning and procedural complications) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 2 (2)
Skin Abrasion (Injury, poisoning and procedural complications) | 3 (3)
Skin Injury (Injury, poisoning and procedural complications) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 10 (10)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 (2)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 3 (3)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Site Bruising (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Vascular Access Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Aortic Bruit (Investigations) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1)
Blood Pressure Increased (Investigations) | 2 (2)
Haemoglobin Decreased (Investigations) | 1 (1)
International Normalised Ratio Abnormal (Investigations) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1)
Nutritional Condition Normal (Investigations) | 1 (1)
Occult Blood (Investigations) | 2 (2)
Occult Blood Positive (Investigations) | 1 (1)
Troponin Increased (Investigations) | 1 (1)
Venous Pressure Jugular Increased (Investigations) | 1 (1)
Vitamin B12 Decreased (Investigations) | 1 (1)
Calcium Deficiency (Metabolism and nutrition disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 2 (2)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Sjogren's Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Myolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Akinesia (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Balance Disorder (Nervous system disorders) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 1 (1)
Cognitive Disorder (Nervous system disorders) | 3 (3)
Corticobasal Degeneration (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 8 (9)
Focal Dyscognitive Seizures (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Hypotonia (Nervous system disorders) | 2 (2)
Migraine (Nervous system disorders) | 3 (3)
Polyneuropathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 6 (6)
Tension Headache (Nervous system disorders) | 1 (1)
Tonic Convulsion (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 4 (4)
Visual Field Defect (Nervous system disorders) | 1 (1)
Device Malfunction (Product Issues) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Psychotic Disorder Due To A General Medical Condition (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5)
Bladder Dilatation (Renal and urinary disorders) | 1 (1)
Calculus Bladder (Renal and urinary disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 6 (6)
Dysuria (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 21 (22)
Nocturia (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1)
Renal Mass (Renal and urinary disorders) | 2 (2)
Urethral Haemorrhage (Renal and urinary disorders) | 1 (1)
Urethral Perforation (Renal and urinary disorders) | 1 (1)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urogenital Haemorrhage (Renal and urinary disorders) | 1 (1)
Adnexa Uteri Mass (Reproductive system and breast disorders) | 1 (1)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (23)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Crusting (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nocturnal Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 3 (3)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 (8)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 (1)
Nail Bed Bleeding (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer Haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Spider Naevus (Skin and subcutaneous tissue disorders) | 1 (1)
Cerumen Removal (Surgical and medical procedures) | 1 (1)
Skin Neoplasm Excision (Surgical and medical procedures) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Extremity Necrosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 6 (6)
Hypertension (Vascular disorders) | 10 (12)
Hypertensive Crisis (Vascular disorders) | 2 (2)
Hypertensive Emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Intermittent Claudication (Vascular disorders) | 2 (2)
Jugular Vein Thrombosis (Vascular disorders) | 1 (1)
Labile Blood Pressure (Vascular disorders) | 2 (2)
Orthostatic Hypotension (Vascular disorders) | 3 (3)
Subclavian Vein Thrombosis (Vascular disorders) | 1 (1)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1)
Varicose Vein Ruptured (Vascular disorders) | 1 (1)
Venous Stenosis (Vascular disorders) | 1 (1)
Venous Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03647475/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03647475/SAP_001.pdf